CLINICAL TRIAL: NCT04609410
Title: Bleeding in Moderate Versus Deep Neuro Muscular Blockade for Laparoscopic Liver Surgery
Brief Title: Bleeding in Laparoscopic Liver Surgery
Acronym: MODELS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MODELS/22/OSR
Record Dates: First submitted 2020-10-09; First posted 2020-10-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Blockade; Intraoperative Bleeding; Hepatic Cancer
Keywords: liver surgery; bleeding; neuromuscular blockade; rocuronium; airway pressure
MeSH Terms: conditions — Blood Loss, Surgical; Liver Neoplasms; Hemorrhage | interventions — Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular blockade (Experimental): During surgery, deep neuromuscular blockade will be achieved with the use of train of four (TOF) monitoring, aiming for a Post-Tetanic Count (PTC) = 0 or PTC = 1 and Train of Four Count (TOFC) = 0. TOF and PTC measurements will be performed every 15 minutes. Boluses of 0,1 mg/kg Rocuronium will be administered if monitored PTC is > 1.
  Complete neuromuscular blockade reversal at the end of surgery will be achieved with an i.v. bolus of Sugammadex (variable dose according to depth of residual blockade) if TOF ratio is ≤ 0.9. If TOF ratio is > 0.9, pharmacological neuromuscular blockade reversal can be avoided.
  Interventions: Procedure: Neuromuscular blockade
- Moderate neuromuscular blockade (Active Comparator): During surgery, a moderate neuromuscular blockade will be achieved with the use of train of four (TOF) monitoring. TOF and Post-Tetanic Count (PTC) measurements will be performed every 15 minutes. Boluses of 0,1 mg/kg Rocuronium will be administered if monitored TOF count is ≥ 1 and/or PTC > 5.
  Complete neuromuscular blockade reversal at the end of surgery will be achieved with an i.v. bolus of Sugammadex (variable dose according to depth of residual blockade) if TOF ratio is ≤ 0.9. If TOF ratio is > 0.9, pharmacological neuromuscular blockade reversal can be avoided.
  Interventions: Procedure: Neuromuscular blockade

INTERVENTIONS:
Procedure: Neuromuscular blockade — Neuromuscular blockade will be achieved via rocuronium intravenous administration and level will be monitored with train of four/post tetanic count monitoring

SUMMARY:
Blood loss during liver resection surgery affects patients morbidity, short and long-term mortality. Among non-surgical interventions to minimize intraoperative blood loss and perioperative blood products transfusion, maintaining conditions of low central venous pressure is considered as standard of care. In animals undergoing laparoscopic hepatectomy, reducing airway pressures represents a minimally invasive measure to reduce central venous pressure and therefore bleeding from the hepatic vein. Neuromuscular blocking agents are usually administered during anesthesia to facilitate endotracheal intubation and to improve surgical conditions: a deep level of neuromuscular blockade has already been shown to reduce peak airway pressures and plateau airway pressures in non-abdominal procedures. Such airway pressures reduction can potentially limit bleeding from hepatic veins during transection phase in liver surgery. The aim of the present study is to evaluate the impact of deep neuromuscular blockade on bleeding (as a consequence of reduced airway peak pressure and plateau pressure) in hepatic laparoscopic resections. Patients undergoing laparoscopic liver resection will be randomized to achieve, using intravenous Rocuronium, either a deep neuromuscular blockade (post-tetanic count = 0 and/or = 1 and train of four count = 0) or moderate neuromuscular blockade (train of four count ≥ 1 and/or post-tetanic count > 5) during surgery. Neuromuscular blockade measurements will be performed every 15 minutes. The primary endpoint is to assess the total blood loss at the end of the resection phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic liver resection
* Patients ≥ 18 years old
* Patients willing to participate to the study and able to validly sign informed consent.

Exclusion Criteria:

* Patients presenting a pre-operative platelet count < 50 x 109/L and/or patients with active pre-operative bleeding
* Patients with planned requirement of continuous neuromuscular blockade monitoring (upon clinical judgement)
* Known hypersensitivity / previous allergic reactions to study medications
* Planned total intra-venous anesthesia technique
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Total intra-operative blood loss | Postoperative day 0
  total blood loss at the end of surgery, measured in milliliters (ml) of blood inside the aspirator canister

SECONDARY OUTCOMES:
Number of blood product units transfused | Up to hospital discharge, an average of 5 days
  number of blood product units transfused from the experimental intervention until hospital discharge
Incidence of surgical revision | Up to hospital discharge, an average of 5 days
  incidence of surgical revision
Airway peak and plateau pressures | Postoperative day 0
  airway pressures, as indicated by ventilator peak pressure (mmHg) and plateau pressure (mmHg) during surgery
Quality of surgical field | Postoperative day 0
  quality of surgical field as assessed by the surgeon with Leiden-Surgical Rating Scale (L-SRS), ranging from 1 (extremely poor conditions) to 5 (optimal conditions), higher scores meaning better outcome
Surgery and hepatic resection time | Postoperative day 0
  surgery and hepatic resection time

OTHER OUTCOMES:
30-day mortality | day 30
  mortality
Pulmonary complications at day 30 | day 30
  rate of pulmonary complications
90-day quality of life | day 90
  quality of life measured with Euro-Quality of Life - 5 Dimensions scale (EQ-5D-5L), composed of:
  * the EQ-5D-5L descriptive system comprising 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension
  * the EQ VAS corresponding to a 20 cm vertical, visual analogue scale ranging from 'the best health you can imagine' to 'the worst health you can imagine'

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zangrillo, Prof., Study Director — IRCCS San Raffaele Scientific Institute; Luigi Beretta, Prof., Study Chair — IRCCS San Raffaele Scientific Institute; Raffaella Reineke, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Background] Ibrahim S, Chen CL, Lin CC, Yang CH, Wang CC, Wang SH, Liu YW, Yong CC, Concejero A, Jawan B, Cheng YF. Intraoperative blood loss is a risk factor for complications in donors after living donor hepatectomy. Liver Transpl. 2006 Jun;12(6):950-7. doi: 10.1002/lt.20746. PMID 16721773
- [Background] Taketomi A, Kitagawa D, Itoh S, Harimoto N, Yamashita Y, Gion T, Shirabe K, Shimada M, Maehara Y. Trends in morbidity and mortality after hepatic resection for hepatocellular carcinoma: an institute's experience with 625 patients. J Am Coll Surg. 2007 Apr;204(4):580-7. doi: 10.1016/j.jamcollsurg.2007.01.035. PMID 17382216
- [Background] Yang T, Zhang J, Lu JH, Yang GS, Wu MC, Yu WF. Risk factors influencing postoperative outcomes of major hepatic resection of hepatocellular carcinoma for patients with underlying liver diseases. World J Surg. 2011 Sep;35(9):2073-82. doi: 10.1007/s00268-011-1161-0. PMID 21656309
- [Background] Moggia E, Rouse B, Simillis C, Li T, Vaughan J, Davidson BR, Gurusamy KS. Methods to decrease blood loss during liver resection: a network meta-analysis. Cochrane Database Syst Rev. 2016 Oct 31;10(10):CD010683. doi: 10.1002/14651858.CD010683.pub3. PMID 27797116
- [Background] Honda G, Kurata M, Okuda Y, Kobayashi S, Tadano S, Yamaguchi T, Matsumoto H, Nakano D, Takahashi K. Totally laparoscopic hepatectomy exposing the major vessels. J Hepatobiliary Pancreat Sci. 2013 Apr;20(4):435-40. doi: 10.1007/s00534-012-0586-7. PMID 23269462
- [Background] Kobayashi S, Honda G, Kurata M, Tadano S, Sakamoto K, Okuda Y, Abe K. An Experimental Study on the Relationship Among Airway Pressure, Pneumoperitoneum Pressure, and Central Venous Pressure in Pure Laparoscopic Hepatectomy. Ann Surg. 2016 Jun;263(6):1159-63. doi: 10.1097/SLA.0000000000001482. PMID 26595124
- [Background] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097
- [Background] Oh SK, Kwon WK, Park S, Ji SG, Kim JH, Park YK, Lee SY, Lim BG. Comparison of Operating Conditions, Postoperative Pain and Recovery, and Overall Satisfaction of Surgeons with Deep vs. No Neuromuscular Blockade for Spinal Surgery under General Anesthesia: A Prospective Randomized Controlled Trial. J Clin Med. 2019 Apr 12;8(4):498. doi: 10.3390/jcm8040498. PMID 31013693